CLINICAL TRIAL: NCT02041299
Title: The Efficacy and Safety of Ferriprox® for the Treatment of Transfusional Iron Overload in Patients With Sickle Cell Disease or Other Anemias
Brief Title: Efficacy and Safety of Ferriprox® in Patients With Sickle Cell Disease or Other Anemias
Acronym: FIRST
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulties with additional recruitment as pool of potential patients was exhausted, and sufficient information for determination of study outcome measure was already obtained
Sponsor: ApoPharma (Industry)
Responsible Party: Sponsor
Organization: Chiesi Canada Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LA38-0411
Record Dates: First submitted 2014-01-15; First posted 2014-01-22 (Estimated); Results first posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-07

CONDITIONS: Iron Overload; Sickle Cell Disease; Other Anemias
Keywords: sickle cell disease; Iron overload; Deferiprone; Ferriprox; deferoxamine; Chelation
MeSH Terms: conditions — Iron Overload; Anemia, Sickle Cell | interventions — Deferiprone; Deferoxamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Deferiprone (Experimental): Patients randomized to the deferiprone arm will be prescribed either tablets or liquid medication. Deferiprone is taken orally, at a dosage that is calculated in terms of milligrams per kilogram of body weight (mg/kg) and is divided into 3 equal doses taken approximately 8 hours apart. The daily dosage is 75 mg/kg (25 mg/kg per dose) for patients with less severe iron load, and 99 mg/kg (33 mg/kg per dose) for those with more severe iron load.
  Interventions: Drug: Deferiprone
- Deferoxamine (Active Comparator): Patients randomized to the deferoxamine arm will be prescribed the drug as per the approved US prescribing information. Deferoxamine is administered as a subcutaneous infusion over 8-12 hours, 5 to 7 days a week. The dosage is 20 mg/kg (children) or 40 mg/kg (adults) in patients with less severe iron load, and up to 40 mg/kg (children) or 50 mg/kg (adults) in those with more severe iron load.
  Interventions: Drug: Deferoxamine

INTERVENTIONS:
Drug: Deferiprone
  Other Names: Ferriprox tablets; Deferiprone oral solution
  Arms: Deferiprone
Drug: Deferoxamine
  Arms: Deferoxamine

SUMMARY:
This research is being done so that we can look at the safety and efficacy of deferiprone in people with sickle cell disease or other anemias. Deferiprone is a drug that removes iron from the body. We will be comparing deferiprone with deferoxamine, another drug that removes iron from the body.

DETAILED DESCRIPTION:
Deferiprone (brand name Ferriprox®) is an iron chelator that is approved in the United States and over 60 other countries for the treatment of iron overload in patients with thalassemia, when other treatments are inadequate. This study has been designed to evaluate the efficacy, safety, and tolerability of deferiprone vs. deferoxamine in patients who have SCD or other anemias, and who require chelation because of the extra iron they are taking in through blood transfusions.

About 300 people from North America, South America, Europe, and the Middle East will take part in this study. Participants will be randomized in a 2:1 ratio to receive therapy for 52 weeks with either deferiprone or deferoxamine, another type of iron chelator. Patients who are randomized to the deferiprone group can choose to get the drug as either tablets or liquid, and must take it three times daily. Patients who are randomized to the deferoxamine group will receive it as a subcutaneous infusion that lasts from 8 to 12 hours and is given 5 to 7 days per week. For both drugs, the starting dosage is based on how much extra iron they have taken in through transfusions in the last 3 months and on the severity of iron load, as measured by serum ferritin levels in the blood and by the amount of iron in the liver and the heart. For deferiprone, the starting dosage will be increased each week over the first 3 weeks; and for both drugs, the dosage may be adjusted up or down during the study based on the level of iron overload and on safety considerations.

Patients will need to have their blood count checked every week for the first 26 weeks, then every other week for the remaining 26 weeks; they will also have to give a blood sample for more detailed safety testing every month; and to give a blood sample for the measurement of serum ferritin every 3 months. Every six months, they will undergo an ECG and an MRI scan, and will be asked to complete a quality of life survey.

At the end of the 52 weeks, participants will be invited to enter a 2-year study in which all patients will receive deferiprone, including those who were randomized to receive deferoxamine in the first year.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 2 years of age;
2. Have sickle cell disease (confirmed by Hb electrophoresis or more specific tests) or other conditions with iron overload from repeated blood transfusions (see exclusion criteria for exceptions);
3. Baseline LIC >7 mg/g dw (measured by MRI);
4. Patients who have received no less than 20 transfusions of RBCs;
5. Patients who have received at least 1 transfusion per year in the last 2 years and who are expected to have a continuing requirement (based on Investigator's judgement) during the duration of the trial

Exclusion Criteria:

1. Thalassemia syndromes;
2. Myelodysplastic syndrome (MDS) or myelofibrosis;
3. Diamond Blackfan anemia;
4. Primary bone marrow failure;
5. Baseline LIC >30 mg/g dw (measured by MRI);
6. Unable or unwilling to undergo a 7 day washout period if currently being treated with deferiprone or deferoxamine or deferasirox;
7. Previous discontinuation of treatment with deferiprone or deferoxamine due to adverse events;
8. History or presence of hypersensitivity or idiosyncratic reaction to deferiprone or deferoxamine;
9. Treated with hydroxyurea within 30 days;
10. History of malignancy;
11. Evidence of abnormal liver function (serum ALT level(s) > 5 times upper limit of normal at screening or creatinine levels >2 times upper limit of normal at screening);
12. A serious, unstable illness, as judged by the Investigator, during the past 3 months before screening/baseline visit including but not limited to: hepatic, renal, gastro-enterologic, respiratory, cardiovascular, endocrinologic, neurologic or immunologic disease;
13. Clinically significant abnormal 12-lead ECG findings;
14. Cardiac MRI T2* <10ms;
15. Myocardial infarction, cardiac arrest or cardiac failure within 1 year before screening/baseline visit;
16. Unable to undergo MRI
17. Presence of metallic objects such as artificial joints, inner ear (cochlear) implants, brain aneurysm clips, pacemakers, and metallic foreign bodies in the eye or other body areas that would prevent use of MRI imaging

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2014-04-17 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2019-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Kwiatkowski, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (33):
- United States (8):
  - Children's Hospital Oakland, Oakland, California
  - University of Illinois at Chicago, Chicago, Illinois
  - Children's Hospital, New Orleans, Louisiana
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - The Children's Hospital of Philadephia, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
- Brazil (5):
  - Centro Infantil Boldrini, Campinas
  - Hospital de Clínicas de Porto Alegre-HCPA,, Rio Branco
  - Instituto Estadual de Hematologia Arthur Siqueira Cavalcanti - HEMORIO, Rio de Janeiro
  - Casa de Saúde Santa Marcelina, São Paulo
  - Universidade Federal de São Paulo, São Paulo
- Hospital for Sick Kids, Toronto, Ontario, Canada
- Egypt (6):
  - Mansoura University Children's Hospital, Al Mansurah
  - Alexandria University, Alexandria
  - Zagazig University, Alexandria
  - Ains Shams University, Cairo
  - Cairo University, Cairo
  - Pediatric Hospital of Cairo University, Cairo
- Saudi Arabia (3):
  - King Abdulaziz University Hospital, Jeddah, Western Region
  - Asser Central Hospital, Abhā
  - King Khalid University Hospital, Riyadh
- Tunisia (3):
  - National Center for Bone Marrow Transplantation, Tunis, Bad Saadoun
  - Farhat Hached Hospital, Hematology Department, Sousse
  - Principal Military Hospital of Instruction of Tunis, Tunis
- Turkey (Türkiye) (3):
  - Cukurova University, Adana
  - Hacettepe University, Ankara
  - Istanbul University, Istanbul
- United Kingdom (4):
  - Hammersmith Hospital, London
  - Barts and The London, London
  - Evelina Children's Hospital, London
  - Imperial College Healthcare NHS Trust, London

REFERENCES:
- [Derived] Kwiatkowski JL, Hamdy M, El-Beshlawy A, Ebeid FSE, Badr M, Alshehri A, Kanter J, Inusa B, Adly AAM, Williams S, Kilinc Y, Lee D, Tricta F, Elalfy MS. Deferiprone vs deferoxamine for transfusional iron overload in SCD and other anemias: a randomized, open-label noninferiority study. Blood Adv. 2022 Feb 22;6(4):1243-1254. doi: 10.1182/bloodadvances.2021004938. PMID 34847228

RESULTS

PARTICIPANT FLOW:
Groups:
- Deferiprone: Patients randomized to the deferiprone arm (daily dosage of either 75 or 99 mg/kg divided into 3 equal doses, taken orally)
- Deferoxamine: Patients randomized to the deferoxamine arm (either 20 mg/kg or up to 40 mg/kg for children, either 40 or 50 mg/kg for adults, administered as a subcutaneous infusion over 8-12 hours, 5 to 7 days a week)
Period: Overall Study
Arm/Group | Deferiprone | Deferoxamine
Started | 152 | 78 (Two participants double-enrolled under different subject numbers so were each counted twice.)
Completed | 106 | 58
Not Completed | 46 | 20
Not completed — Adverse Event | 9 | 3
Not completed — Lost to Follow-up | 4 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 13 | 7
Not completed — Protocol Violation | 11 | 4
Not completed — Termination of the study | 7 | 3
Not completed — Required bone marrow transplant | 0 | 1
Not completed — Patient stopped dosing on unknown date | 1 | 0

BASELINE CHARACTERISTICS:
Population: Number of patients who received study product
Groups:
- Deferiprone: Number of patients who received deferiprone
- Deferoxamine: Number of patients who received deferoxamine
- Total: Total of all reporting groups
Arm/Group | Deferiprone | Deferoxamine | Total
Number analyzed (Participants) | 152 | 76 | 228
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.9 (10.2) | 16.9 (8.5) | 16.9 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 38 | 107
  Male | 83 | 38 | 121
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 6 | 16
  Not Hispanic or Latino | 142 | 70 | 212
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 23 | 14 | 37
  White | 120 | 56 | 176
  More than one race | 9 | 6 | 15
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Saudi Arabia | 8 | 3 | 11
  Canada | 1 | 1 | 2
  Turkey | 1 | 1 | 2
  United States | 16 | 7 | 23
  Egypt | 105 | 51 | 156
  Brazil | 9 | 7 | 16
  United Kingdom | 6 | 5 | 11
  Tunisia | 6 | 1 | 7
Liver iron concentration at baseline [Mean (Standard Deviation); unit: mg iron per gram of liver dry weight] — Liver iron concentration (LIC), measured by MRI as milligrams of iron per gram of liver dry weight. A value > 7 mg/g dw is indicative of iron overload.
  mg iron per gram of liver dry weight | 16.54 (7.49) | 15.97 (7.20) | 16.26 (7.30)
Cardiac iron at baseline [Mean (Standard Deviation); unit: milliseconds] | 33.52 (6.26) | 33.87 (6.17) | 33.64 (6.22)
Serum ferritin level at baseline [Mean (Standard Deviation); unit: micrograms per liter] | 4125.4 (2407.4) | 4055.3 (2708.5) | 4101.89 (2505.66)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Liver Iron Concentration (LIC)
Description: LIC was measured by MRI. A score >7 mg/g dw is indicative of iron overload.
Time Frame: Change from baseline to Week 52
Population: Intent-to-treat population
Measure: Least Squares Mean (Standard Error); unit: mg of iron per gram of liver dry weight
Groups:
- Deferiprone: Patients who received deferiprone and were evaluable for LIC and cardiac MRI T2*
- Deferoxamine: Patients who received deferoxamine and were evaluable for LIC and cardiac MRI T2*
Arm/Group | Deferiprone | Deferoxamine
Number analyzed (Participants) | 122 | 63
mg of iron per gram of liver dry weight | -4.13 (0.50) | -4.38 (0.59)
Statistical Analysis 1: Comparison: Deferiprone vs Deferoxamine; Test type: Non-Inferiority — Non-inferiority is demonstrated if the upper limit of the 96.01% confidence interval (CI) is less than or equal to 2 mg/g dw; p = 0.0399, ANCOVA; Mean Difference (Net) = 0.26, 96.01% CI 2-sided [-0.97 to 1.48]

2. Secondary Outcome: Change From Baseline in Cardiac Iron
Description: Cardiac iron is measured by MRI in milliseconds (ms). A score of less than 20 ms is indicative of cardiac iron overload.
Time Frame: Change from baseline to Week 52
Population: Intent-to-treat population
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Arm/Group | Deferiprone | Deferoxamine
Number analyzed (Participants) | 122 | 63
milliseconds | -0.022068 (0.021133) | -0.021773 (0.025261)
Statistical Analysis 1: Comparison: Deferiprone vs Deferoxamine; Data for this measure were log-transformed; Test type: Non-Inferiority — Support for non-inferiority is demonstrated if the 96.01% CI contains zero (0); p = 0.0399, ANCOVA; Mean Difference (Net) = -0.000295, 96.01% CI 2-sided [-0.054247 to 0.053657]

3. Secondary Outcome: Change From Baseline in Serum Ferritin
Description: Serum ferritin provides a measure of iron level in the blood. Normal levels of serum ferritin are under 300 µg/L for females and 400 µg/L for males.
Time Frame: Change from baseline to Week 52
Population: Intent-to-treat
Measure: Least Squares Mean (Standard Error); unit: micrograms per liter
Groups:
- Deferiprone: Patients who received deferiprone and were evaluable for serum ferritin. In contrast to liver and cardiac iron, for which the first post-baseline assessment took place at Month 6, that for serum ferritin took place at Month 3. Since fewer patients had withdrawn by Month 3 than by Month 6, there were more evaluable patients for this measure than for the other two.
- Deferoxamine: Patients who received deferoxamine and were evaluable for serum ferritin. In contrast to liver and cardiac iron, for which the first post-baseline assessment took place at Month 6, that for serum ferritin took place at Month 3. Since fewer patients had withdrawn by Month 3 than by Month 6, there were more evaluable patients for this measure than for the other two.
Arm/Group | Deferiprone | Deferoxamine
Number analyzed (Participants) | 133 | 67
micrograms per liter | -385.83 (234.05) | -760.89 (289.40)
Statistical Analysis 1: Comparison: Deferiprone vs Deferoxamine; Test type: Non-Inferiority — Support for non-inferiority of deferiprone to deferoxamine in serum ferritin is demonstrated if the 96.01% CI contains zero (0); p = 0.0399, ANCOVA; Mean Difference (Net) = 375.07, 96.01% CI 2-sided [-260.63 to 1010.76]

4. Secondary Outcome: Change in Patient-reported Quality of Life, as Measured by the Short Form Health Survey (SF-36) or the Child Health Questionnaire (CHQ-PF50).
Description: Adult patients completed the SF-36 questionnaire and minors completed the CHQ-PF50. These questionnaires yield a profile of functional health and well-being, based on 8 scales of physical and mental health measures: Physical Functioning, Role Limitations due to Physical Health, Bodily Pain, General Health Perceptions, Vitality, Social Functioning, Role Limitations due to Emotional Problems, and Mental Health (MH), and summary scores are produced for physical well-being and mental well-being. The summaries are scored from 0-100, with higher scores reflecting better outcomes.
Time Frame: Change from baseline to Week 52
Population: Due to administrative and other issues, a majority of participants were missing scores. Evaluable data were obtained from 35 DFP and 19 DFO patients for the SF-36, and from 60 DFP and 23 DFO patients for the CHQ.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Deferiprone: Patients who received deferiprone and were evaluable for quality of life
- Deferoxamine: Patients who received deferoxamine and were evaluable for quality of life
Arm/Group | Deferiprone | Deferoxamine
Number analyzed (Participants) | 95 | 42
score on a scale
  SF-36 Physical Summary: number analyzed (Participants) | 35 | 19
  SF-36 Physical Summary | 43.1 (1.8) | 43.0 (2.0)
  SF-36 Mental Summary: number analyzed (Participants) | 35 | 19
  SF-36 Mental Summary | 44.7 (2.7) | 40.9 (2.9)
  CHQ-PF50 Physical Summary: number analyzed (Participants) | 60 | 23
  CHQ-PF50 Physical Summary | 29.3 (1.8) | 30.5 (2.4)
  CHQ-PF50 Psychosocial Summary: number analyzed (Participants) | 60 | 23
  CHQ-PF50 Psychosocial Summary | 42.5 (1.5) | 41.3 (2.1)
Statistical Analysis 1: Comparison: Deferiprone vs Deferoxamine; Test type: Superiority — Comparison of treatment groups on change in score on SF-36 Physical Summary; p = 0.9214, ANCOVA
Statistical Analysis 2: Comparison: Deferiprone vs Deferoxamine; Comparison of treatment groups on change in score on SF-36 Mental Summary; Test type: Superiority; p = 0.1174, ANCOVA
Statistical Analysis 3: Comparison: Deferiprone vs Deferoxamine; Comparison of treatment groups on change in score on CHQ-PF50 Physical Summary; Test type: Superiority; p = 0.6488, ANCOVA
Statistical Analysis 4: Comparison: Deferiprone vs Deferoxamine; Comparison of treatment groups on change in score on CHQ-PF50 Psychosocial Summary; Test type: Superiority; p = 0.5915, ANCOVA

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Deferiprone: Patients randomized to the deferiprone arm will be prescribed either tablets or liquid medication.
  Deferiprone
- Deferoxamine: Patients randomized to the deferoxamine arm will be prescribed the drug as per the approved US prescribing information.
  Deferoxamine
Arm/Group | Deferiprone | Deferoxamine
All-Cause Mortality (participants affected / at risk) | 1/152 | 1/76
Serious Adverse Events (participants affected / at risk) | 40/152 | 14/76
Other Adverse Events (participants affected / at risk) | 134/152 | 67/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deferiprone (N=152) | Deferoxamine (N=76)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypersplenism (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 4 (5) | 1 (2)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 16 (31) | 4 (8)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal pain/upper (Gastrointestinal disorders) | 3 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Malaise (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 5 (5) | 3 (5)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic sequestration (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis fulminant (Hepatobiliary disorders) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1)
Parvovirus infection (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 2 (3)
Propionibacterium infection (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vascular device infection (Infections and infestations) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Transaminases increased (Investigations) | 2 (2) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Bone infarction (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Hip surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Splenectomy (Surgical and medical procedures) | 2 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deferiprone (N=152) | Deferoxamine (N=76)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 21 (57) | 9 (17)
Abdominal pain/upper (Gastrointestinal disorders) | 37 (86) | 10 (13)
Diarrhoea (Gastrointestinal disorders) | 6 (8) | 5 (10)
Nausea (Gastrointestinal disorders) | 11 (14) | 6 (6)
Toothache (Gastrointestinal disorders) | 3 (3) | 5 (5)
Vomiting (Gastrointestinal disorders) | 28 (59) | 7 (8)
Chest pain (General disorders) | 5 (6) | 4 (4)
Injection site pain (General disorders) | 0 (0) | 5 (6)
Injection site swelling (General disorders) | 0 (0) | 4 (8)
Pain (General disorders) | 8 (13) | 3 (3)
Pyrexia (General disorders) | 40 (65) | 22 (33)
Influenza (Infections and infestations) | 5 (8) | 5 (5)
Nasopharyngitis (Infections and infestations) | 14 (22) | 9 (13)
Alanine aminotransferase increased (Investigations) | 18 (27) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 17 (26) | 0 (0)
Neutrophil count decreased (Investigations) | 12 (16) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (24) | 6 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 20 (33) | 13 (25)
Bone pain (Musculoskeletal and connective tissue disorders) | 38 (92) | 26 (62)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 (36) | 11 (15)
Headache (Nervous system disorders) | 30 (54) | 10 (17)
Chromaturia (Renal and urinary disorders) | 9 (10) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 11 (13)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 15 (19) | 11 (13)

LIMITATIONS AND CAVEATS:
The trial was terminated early as the pool of potential participants was exhausted and it was determined that the number of patients already randomized would be sufficient to assess the primary endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-05-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT02041299/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-03): https://cdn.clinicaltrials.gov/large-docs/99/NCT02041299/SAP_001.pdf